CLINICAL TRIAL: NCT02831959
Title: Pivotal, Open-label, Randomized Study of Radiosurgery With or Without Tumor Treating Fields (TTFields) for 1-10 Brain Metastases From Non-small Cell Lung Cancer (NSCLC).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-25 METIS
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases From Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer; NSCLC; Brain metastases; Treatment; Minimal toxicity; TTFields; TTF; Tumor Treating Fields; Novocure; SRS; Stereotactic radiosurgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NovoTTF-200M device (Experimental): NovoTTF-200M device Patients undergo SRS followed by continuous TTFields treatment using the NovoTTF-200M device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the head.
  The treatment enables the patient to maintain regular daily routine.
  Interventions: Device: NovoTTF-200M device; Other: Best Standard of Care
- Best Standard of Care (Active Comparator): Patients will undergo SRS alone and be treated with the best known standard of care for Non-Small Cell Lung Cancer metastatic to the brain.
  Interventions: Other: Best Standard of Care

INTERVENTIONS:
Device: NovoTTF-200M device
  Arms: NovoTTF-200M device
Other: Best Standard of Care

SUMMARY:
The study is a prospective, randomized controlled phase III trial, to test the efficacy, safety and neurocognitive outcomes of advanced NSCLC patients, following stereotactic radiosurgery (SRS) for 1 inoperable brain metastasis or 2-10 brain metastases, treated with NovoTTF-200M and supportive treatment compared to supportive treatment alone. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo NSCLC pre-clinical models both as a single modality treatment and in combination with chemotherapies. TTFields have also shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a pilot study, 42 patients with advanced NSCLC who had tumor progression after at least one line of prior chemotherapy, received pemetrexed together with TTFields (150 kHz) applied to the chest and upper abdomen until disease progression (Pless M., et al., Lung Cancer 2011). Efficacy endpoints were remarkably high compared to historical data for pemetrexed alone.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate) (Stupp R., et al., EJC 2012). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life (Stupp R., et al., JAMA 2015).

Applying TTFields at 150 kHz to the brain for the treatment of 1-5 brain metastasis from NSCLC using the NovoTTF-100M device has been demonstrated to be safe in a pilot study, where patients were randomized after local therapy of their brain metastasis by neurosurgery and/or stereotactic radiosurgery to receive either NovoTTF-100M treatment or supportive care alone. Eighteen (18) patients have been enrolled in the study. There have been no device-related serious adverse events (SAE) reported to date (Brozova H., et al., Neuro Oncol 2016).

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with 1-10 brain metastases from NSCLC which are amenable to stereotactic radiosurgery (SRS). In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

1. Patients undergo SRS followed by TTFields using the NovoTTF-200M System
2. Patients undergo SRS alone and receive supportive care. Patients in both arms of the study may receive systemic therapy for their NSCLC at the discretion of their treating physician.

Patients will be randomized at a 1:1 ratio. Baseline tests will be performed in patients enrolled in both arms. If assigned to the NovoTTF-200M group, the patients will be treated continuously with the device until second intracranial progression.

On both arms, patients who recur anywhere in the brain will be offered one of the following salvage treatments (according to local practice) including, but not limited to:

* Surgery
* Repeat SRS
* Whole brain radiotherapy (WBRT) Patients on the control arm will be offered to cross over to the NovoTTF-200M arm of the study and receive TTFields with or without salvage therapy for second intracranial progression if the investigator believes it is in the best interest of the patient and patient agrees.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically- charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death.. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues. In conclusion, TTFields hold the promise of serving as a brand new treatment for brain metastases from NSCLC with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Life expectancy of ≥ 3 months
3. New diagnosis of brain metastases from a histologically or cytologically confirmed primary or metastatic NSCLC tumor within 5 years of registration on the study. If the original histological proof of malignancy is greater than 5 years, then pathological confirmation is required (i.e.: from extra-cranial or intracranial disease).

5. 1 inoperable brain metastasis or 2- 10 brain lesions per screening MRI, confirmed by contrast enhanced MRI amenable to SRS according to the following criteria:

a. largest tumor volume < 10 cc b. longest tumor diameter < 3 cm c. Cumulative volume of all tumors ≤ 15 cc 6. At least one measurable disease per study protocol 7. Patients must be receiving optimal therapy for their extracranial disease according to local practice at each center. Patients may continue on systemic therapy while receiving TTFields.

8. Able to operate the NovoTTF-200M device independently or with the help of a caregiver 9. Clinical trials prior to enrollment are allowed, as long as no brain directed therapy was included (current treatment trials are exclusionary)

Exclusion Criteria:

1. Patients who are known to have somatic tumor mutations in the following genes, for which targeted agents are available that directly affect the treatment of brain metastasis: Anaplastic lymphoma kinase (ALK), epidermal growth factor receptor (EGFR), ROS-1 proto- oncogene, and proto-oncogene B-RAF
2. Patients who have a single, operable brain metastasis
3. Patients with significant edema leading to risk of brain herniation
4. Patients with midline shift > 10mm
5. Patients with intractable seizures
6. Leptomeningeal metastases
7. Recurrent brain metastases
8. Prior WBRT for newly diagnosed brain metastases
9. Severe comorbidities:

   1. Clinically-significant inadequate hematological, hepatic and renal function, defined as: Neutrophil count < 1.5 x 10 9/L and platelet count < 100 x 10^9/L; bilirubin > 1.5 x upper limit of normal (ULN); aspartate transaminase (AST) and/or alanine aminotransferase (ALT) > 2.5 x ULN or > 5 x ULN if patient has documented liver metastases; and serum creatinine > 1.5 x ULN
   2. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/ third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea).
   3. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the study.
   4. History of cerebrovascular accident (CVA) within 6 months prior to randomization or that is not stable
   5. Active infection or serious underlying medical condition that would impair the ability of the patient to received protocol therapy
   6. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
10. Implantable electronic medical devices in the brain
11. Known allergies to medical adhesives or hydrogel
12. Currently pregnant or breastfeeding
13. Planned concurrent brain directed therapy (beyond SRS and NovoTTF-200M as per protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-07; Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Time to intracranial progression | 3 years

SECONDARY OUTCOMES:
Time to neurocognitive failure | 3 years
  Measured by cognitive decline on a battery of tests: Hopkins Verbal Learning Test (HVLT-R) free recall, delayed recall, and delayed recognition; Controlled Oral Word Association Test (COWAT); and Trail Making Tests (TMT) Parts A and B
Overall survival | 3 years
Radiological response in the brain following study treatments | 3 years
Time to second intracranial progression | 3 years
Time to intracranial progression, measured from the date of first SRS treatment to intracranial progression (per modified RECIST 1.1 Criteria) or neurological death, whichever occurs first. | 3 years
Time to first and second intracranial progression evaluated in two cohorts of patients, 1-4 brain metastases and 5-10 brain metastases. | 3 years
Rate of intracranial progression at 2, 4, 6, 8, 10, 12 months after first SRS treatment | 3 years
Time to distant progression, as measured from the date of first SRS treatment to a new intracranial lesion | 3 years
Rate of decline in cognitive function as measured by HVLT-R free recall, delayed recall and delayed recognition, COWAT and TMT Parts A and B at 2, 4, 6, 8, 10, 12 months follow-up. | 3 years
Neurocognitive failure-free survival | 3 years
  Defined from the date of first SRS treatment to neurocognitive failure (as measured by HVLT-R free recall, delayed recall, and delayed recognition; COWAT; and TMT Parts A and B) or death (whichever occurs first), censored at the last neurocognitive assessment on which the patient was reported alive without neurocognitive failure
Quality of Life using the EORTC QLQ C30 with BN20 addendum | 3 years
Toxicity during NovoTTF-200M treatment based on incidence and severity of treatment emergent adverse events as evaluated using the CTCAE version 4.0 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Minesh Mehta, MD, Principal Investigator — Miami Cancer Institute, Miami FL USA; Paul Brown, MD, Principal Investigator — MD Anderson Cancer Center, Houston TX USA; Vinai Gondi, MD, Principal Investigator — Northwestern Medicine Cancer Center, Warenville IL USA; Manmeet Ahluwalia, MD, Principal Investigator — Cleveland Clinic, Cleveland OH USA
Locations (128):
- United States (61):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Grandview Medical Center - Cancer Center, Birmingham, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - MemorialCare Cancer Institute, Long Beach, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - Kaiser Permanente Redwood City, Redwood City, California
  - Dignity Health - Mercy Cancer Centers, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Sharp HealthCare, San Diego, California
  - University of California, San Francisco, California
  - St. Mary's Medical Center - Grand Junction, Grand Junction, Colorado
  - Banner North Colorado Medical Center (NCMC) - Oncology - Greeley, Greeley, Colorado
  - Banner MD Anderson Cancer Center - McKee Medical Center, Loveland, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Adult Oncology Research, Orlando, Florida
  - UF Health Cancer Center, Orlando, Florida
  - BRCR Medical Center INC, Plantation, Florida
  - Piedmont Brain Tumor Center, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - CDH-Delnor Health System, Warrenville, Illinois
  - University of Kansas Cancer Center and Medical Pavilion, Kansas City, Kansas
  - University of Kentucky HealthCare, Lexington, Kentucky
  - University of Louisville-James Graham Brown Cancer Center, Louisville, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Abbott Northwestern Hospital - Givens Brain Tumor Center, Minneapolis, Minnesota
  - John Nasseff Neuroscience Institute ANW Brain Tumor Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center (UMMC) - Fairview - Masonic Cancer Clinic, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, University of Missouri Healthcare, Columbia, Missouri
  - Oncology Research | Mercy Research, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - UNC - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina- Hollings Cancer Center, Charleston, South Carolina
  - Prisma Health - Upstate, Greenville, South Carolina
  - Erlanger Baroness Hospital, Chattanooga, Tennessee
  - West Cancer Center, Germantown, Tennessee
  - Mischer Neuroscience Associates - Texas Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Oncology, McKinney, Texas
  - Texas Oncology, Plano, Texas
  - Baylor Scott & White Medical Center - Temple, Waco, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Bulgaria (2):
  - UMHAT Sv. Ivan Rilski EAD, Department of Medical Oncology, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed, Department of Medical Oncology, Sofia
- Canada (5):
  - Cancercare Manitoba, Winnipeg, Manitoba
  - Le CIUSSS de I'Est-de-L'ile de Montreal - Hôpital Maisonneuve Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - (CHUS) Centre Hospitalier Universitaire de Sherbrooke, Service de Neurochirurgie, Sherbrooke, Quebec
- China (22):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Chaoyang
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Xuhui District
  - Taizhou Hospital, Zhejiang Province, Zhejiang, Zhejiang
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Affiliated Hospital Of Xingtai Medical College, Hebei
  - The First Hospital of China Medical University, Shenyang
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - The First Affiliated Hospital of Xiamen University, Xiamen
- Radiochirugia Zagreb, Sveta Nedelja, Croatia
- France (4):
  - University Hospital Lille, Lille
  - Clairval Hospital Center, Marseille
  - Hopital Pitié-Salpétriere, Paris
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Etienne
- Germany (6):
  - Klinik für Radioonkologie und Strahlentherapie der Charité Universitätsmedizin Berlin Campus Charité Virchow-Klinikum, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Dr. Senckenbergisches Institut for Neurooncology,, Frankfurt am Main
  - Dr. Senckenbergisches Institut für Neuroonkologie, Zentrum der Neurologie und Neurochirurgie, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Klinik für Innere Medizin IV, Hämatologie / Onkologie, Halle
  - Heidelberg University Clinic for Radiooncology and Radiation Therapy, Heidelberg
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - National Koranyi Institute of Tb and Pulmonology, Budapest
  - Onkologiai Osztaly, Balassa Janos Korhaz, Szekszárd
  - Geza Hetenyi Hospital-Clinic of Jasz-Nagykun-Szolnok County, Szolnok
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (7):
  - A.O.S.G. Moscati Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialità, Avellino
  - General Hospital Gavazzeni, Bergamo
  - Radioterapia Oncologica AOU Careggi, Florence
  - Azienda Socio Sanitaria Territoriale di Lecco, Lecco
  - University Hospital of Messina AOU Policlinico "G. Martino", Messina
  - The IRCCS Carlo Besta Neurological Institute Foundation, Milan
  - A.O.U Città della Salute e della Scienza di Torino, Torino
- Poland (6):
  - Marek Harat Private Practice, Neurosurgery and Radiation Oncology, Bydgoszcz
  - University Clinical Center, Gdansk
  - Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice
  - MS Clinsearch Sp. z.o.o., Lublin
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Gamma Knife Center Warsaw, Warsaw
- Center for Neuro-oncology, Neurosurgery Clinic, Clinical Center of Serbia, Belgrade, Serbia
- Spain (3):
  - Catalan Institute of Oncology, Barcelona
  - Hospital Universitario HM Sanchinarro Edificio CIOCC, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Giladi M, Weinberg U, Schneiderman RS, Porat Y, Munster M, Voloshin T, Blatt R, Cahal S, Itzhaki A, Onn A, Kirson ED, Palti Y. Alternating electric fields (tumor-treating fields therapy) can improve chemotherapy treatment efficacy in non-small cell lung cancer both in vitro and in vivo. Semin Oncol. 2014 Oct;41 Suppl 6:S35-41. doi: 10.1053/j.seminoncol.2014.09.006. Epub 2014 Sep 8. PMID 25213867
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Brozova H, Lucas A, Salmaggi A, Vymazal J. COMET: A phase II randomized study of TTFields versus supportive care in non-small cell lung cancer patients with 1-5 brain metastases - initial safety results. Neuro Oncol. 2015 Nov; 17 (suppl 5): v46. doi:10.1093/neuonc/nov208.6